CLINICAL TRIAL: NCT05859854
Title: Cenobamate in Adults With Focal-Onset Seizures: a Real-World Multicenter Observational Italian
Brief Title: Cenobamate in Adults With Focal-Onset Seizures
Acronym: BLESS
Status: Active, not recruiting | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 153(A)IM21348
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy; Focal-Onset Seizure; Neurological Disorder
Keywords: cenobamate; Real-word; epilepsy; focal-onset seizure; observational; focal epilepsy uncontrolled
MeSH Terms: conditions — Epilepsy; Seizures; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients diagnosed treated with adjunctive cenobamate in Italy.: Adult patients diagnosed with focal epilepsy uncontrolled despite the use of at least two antiepileptic medicinal products, treated with adjunctive cenobamate in Italy.
  A single cohort of patients will be involved in the study, enrolling both subjects who initiated cenobamate treatment in accordance with the current clinical practice, and subjects previously included in the cenobamate Compassionate Use Programme in Italy, provided that they fulfil all of the eligibility criteria listed below

SUMMARY:
The BLESS Study contributes to filling this information gap by collecting data from the Italian clinical practice and the Compassionate Use Program, to better characterize the clinical profile of cenobamate describing its effectiveness, safety and tolerability in adult patients diagnosed with uncontrolled focal epilepsy despite the use of at least two antiepileptic medicinal products.

DETAILED DESCRIPTION:
The main objective of the study is to describe the effectiveness of adjunctive cenobamate treatment in adult patients with uncontrolled focal epilepsy in Italy, overall and according to age class, setting of cenobamate treatment, cenobamate final target daily dose prescribed, and number of concomitant Anti Seizure Medications (ASMs). This will be assessed by intra-patient percent change and achievement of a ≥50% reduction in the seizure frequency from the pre-treatment baseline over a period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of cenobamate treatment initiation
* Male or female patients
* Patients diagnosed with focal epilepsy uncontrolled despite a history of treatment with at least two antiepileptic medicinal products at the time of cenobamate treatment initiation in agreement with the Summary of Product Characteristics (SmPC)
* Patients who at enrolment had received at least 12 weeks (titration period up to the initial recommended target dose of 200 mg daily completed) but no more than 52 weeks of cenobamate as adjunctive treatment of focal-onset seizures with or without secondary generalization
* Patients with available retrospective data in medical charts and seizure diaries, including information about baseline seizure frequency prior to cenobamate treatment initiation
* Patients who gave written informed consent to take part into the study and personal data processing consent following local regulation.
* Patients who received adjunctive cenobamate for at least 12 weeks and discontinued permanently treatment before enrolment will also be included in the study-

Exclusion Criteria:

* Patients diagnosed with familial short-QT syndrome
* Patients affected by hypersensitivity to the active substance cenobamate or to any of the excipients (e.g., lactose monohydrate)
* Patients with history of severe drug-induced hypersensitivity reaction, including (but not limited to) drug reaction with eosinophilia and systemic symptoms (DRESS), and Stevens Johnson syndrome
* Patients enrolled in a clinical trial in which treatments for epilepsy are managed through a study protocol
* Patient unable to read and write in Italian language and to autonomously fill in questionnaires and scales
* Patients with a known pregnancy or who are breast-feeding from cenobamate treatment initiation till enrolment visit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with focal epilepsy uncontrolled despite the use of at least two antiepileptic medicinal products, treated with adjunctive cenobamate in Italy. A single cohort of patients will be involved in the study, enrolling both subjects who initiated cenobamate treatment in accordance with the current clinical practice, and subjects previously included in the cenobamate Compassionate Use Programme in Italy, provided that they fulfil all of the eligibility criteria listed below
Sampling Method: Probability Sample
Enrollment: 936 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Absolute frequency of patients achieving a 50 % or greater reduction in the seizure frequency (overall) | 12, 24 and 52 weeks of cenobamate treatment initiation
  Seizure frequency during the baseline and post-baseline assessments was calculated by summing the total number of seizures (all types of seizures) reported in each considered period and dividing by the duration of that period (number of days), excluding days with no available diary data, and multiplying by 28 to normalize to a monthly rate ("monthly seizure frequency").
Relative frequency of patients achieving a ≥50% (50% or greater) reduction in the seizure frequency (overall) | 12, 24 and 52 weeks of cenobamate treatment initiation
  Seizure frequency during the baseline and post-baseline assessments was calculated by summing the total number of seizures (all types of seizures) reported in each considered period and dividing by the duration of that period (number of days), excluding days with no available diary data, and multiplying by 28 to normalize to a monthly rate ("monthly seizure frequency").
Intra-patient percent change in the seizure frequency (overall) | 12, 24 and 52 weeks of cenobamate treatment initiation
  Intra-patient percent change from baseline will be defined as [(monthly seizure frequency at post-baseline assessments - monthly seizure frequency at baseline), divided by the monthly seizure frequency at baseline] multiplied by 100.
Absolute frequency of patients achieving a 50 % or greater reduction in the seizure (stratified) | 12, 24 and 52 weeks of cenobamate treatment initiation
  Seizure frequency during the baseline and post-baseline assessments was calculated by summing the total number of seizures (all types of seizures) reported in each considered period and dividing by the duration of that period (number of days), excluding days with no available diary data, and multiplying by 28 to normalize to a monthly rate ("monthly seizure frequency").
  Population will be stratified according to the following:
  * Age class of patient at the time of cenobamate treatment initiation (i.e., <65 years; ≥65 years).
  * Setting of cenobamate treatment initiation (i.e., CUP; current clinical practice).
  * Cenobamate final target daily dose prescribed (i.e., 200 mg; >200 mg).
  * Number of ASMs concomitant with cenobamate (i.e., ≤2 ASMs; >2 ASMs).
Relative frequency of patients achieving a ≥50% (50% or greater) reduction in the seizure frequency (stratified) | 12, 24 and 52 weeks of cenobamate treatment initiation
  Seizure frequency during the baseline and post-baseline assessments was calculated by summing the total number of seizures (all types of seizures) reported in each considered period and dividing by the duration of that period (number of days), excluding days with no available diary data, and multiplying by 28 to normalize to a monthly rate ("monthly seizure frequency").
  Population will be stratified according to the following:
  * Age class of patient at the time of cenobamate treatment initiation (i.e., <65 years; ≥65 years).
  * Setting of cenobamate treatment initiation (i.e., CUP; current clinical practice).
  * Cenobamate final target daily dose prescribed (i.e., 200 mg; >200 mg).
  * Number of ASMs concomitant with cenobamate (i.e., ≤2 ASMs; >2 ASMs).
Intra-patient percent change in the seizure frequency (stratified) | 12, 24 and 52 weeks of cenobamate treatment initiation
  Intra-patient percent change from baseline will be defined as [(monthly seizure frequency at post-baseline assessments - monthly seizure frequency at baseline), divided by the monthly seizure frequency at baseline] multiplied by 100.
  Population will be stratified according to the following:
  * Age class of patient at the time of cenobamate treatment initiation (i.e., <65 years; ≥65 years).
  * Setting of cenobamate treatment initiation (i.e., CUP; current clinical practice).
  * Cenobamate final target daily dose prescribed (i.e., 200 mg; >200 mg).
  * Number of ASMs concomitant with cenobamate (i.e., ≤2 ASMs; >2 ASMs).

SECONDARY OUTCOMES:
Absolute frequency of patients achieving a ≥50%/≥75%/≥90%/=100% sustained reduction in the seizure frequency | 24 and 52 weeks of cenobamate treatment initiation.
  Sustained seizure frequency reduction will be defined as a ≥50%/≥75%/≥90%/=100% reduction in baseline seizure frequency achieved at 12 weeks of cenobamate treatment initiation, that continues (is sustained) without interruption and without cenobamate permanent discontinuation through the observation period until 24 and 52 weeks of cenobamate treatment initiation, respectively.
Absolute frequency of patients achieving a ≥75%/≥90%/=100% reduction in the seizure frequency | 12, 24 and 52 weeks of cenobamate treatment initiation.
  Seizure frequency reduction will be defined as a ≥75%/≥90%/=100% reduction in baseline seizure frequency achieved at 12, 24 and 52 weeks of cenobamate treatment initiation, respectively.
Relative frequencies of patients achieving a ≥50%/≥75%/≥90%/=100% sustained reduction in the seizure frequency | 24 and 52 weeks of cenobamate treatment initiation.
  Sustained seizure frequency reduction will be defined as a ≥50%/≥75%/≥90%/=100% reduction in baseline seizure frequency achieved at 12 weeks of cenobamate treatment initiation, that continues (is sustained) without interruption and without cenobamate permanent discontinuation through the observation period until 24 and 52 weeks of cenobamate treatment initiation, respectively
Relative frequencies of patients achieving a ≥75%/≥90%/=100% reduction in the seizure frequency | 12, 24 and 52 weeks of cenobamate treatment initiation.
  Seizure frequency reduction will be defined as a ≥75%/≥90%/=100% reduction in baseline seizure frequency achieved at 12, 24 and 52 weeks of cenobamate treatment initiation.
Absolute frequency of patients with at least one AE | Through study completion, an average of 1 year
  Absolute frequency of patients treated with cenobamate who experienced at least one AE during the applicable observation period
Relative frequency of patients with at least one AE | Through study completion, an average of 1 year
  Relative frequency of patients treated with cenobamate who experienced at least one AE during the applicable observation period
Absolute frequency of patients with at least one ADR | Through study completion, an average of 1 year
  Absolute frequency of patients treated with cenobamate who experienced at least one ADR during the applicable observation period
Relative frequency of patients with at least one ADR | Through study completion, an average of 1 year
  Relative frequency of patients treated with cenobamate who experienced at least one ADR during the applicable observation period
Absolute frequency of patients treated with at least one SAE | Through study completion, an average of 1 year
  Absolute frequency of patients treated with at least one SAE during the applicable observation period
Relative frequency of patients treated with at least one SAE | Through study completion, an average of 1 year
  Relative frequency of patients treated with at least one SAE during the applicable observation period
Health-Related Quality of life (HRQoL) | 12, 24 and 52 weeks
  The Health-Related Quality of life (HRQoL) of patients will be assessed by means of the 31-item Quality Of Life In Epilepsy inventory (QOLIE-31).
  The 31-item Quality Of Life In Epilepsy inventory (QOLIE-31) is a patient self-reported instrument that contains 31 items grouped in seven multi-item scales ( "seizure worry", "overall QoL", "emotional well-being", "energy fatigue", "cognitive functioning", "medication effects" and "social functioning"). Different items in the QOLIE-31 have different ranges of precoded numeric values, so the scoring procedure requires conversion from raw, precoded numeric values to scores of 0-100 points, with higher scores reflecting better quality of life. The QOLIE-31 overall score is calculated by summing the product of each scale score times its weight and summing over all scales, according to the instructions obtained from copyright holders.
Patient Global functioning (CGI-S) | 12, 24 and 52 weeks
  The patient global functioning will be assessed by means of the Clinical Global Impression (CGI) Scales. The Early Clinical Drug Evaluation Program (ECDEU) version of the CGI is a 3-item clinician rated scale that measures illness severity (CGI-S), global improvement or change (CGI-I) and treatment response (efficacy index: CGI-E).
  The CGI-S score ranges from 1 (normal) through to 7 (amongst the most severely ill patients).
  The calculation of the scores will be performed according to the instructions obtained from copyright holders.
Patient Global functioning (CGI-I) | 12, 24 and 52 weeks
  The patient global functioning will be assessed by means of the Clinical Global Impression (CGI) Scales. The Early Clinical Drug Evaluation Program (ECDEU) version of the CGI is a 3-item clinician rated scale that measures illness severity (CGI-S), global improvement or change (CGI-I) and treatment response (efficacy index: CGI-E).
  The CGI-I score ranges from 1 (very much improved) through to 7 (very much worse).
  The calculation of the scores will be performed according to the instructions obtained from copyright holders.
Patient Global functioning (CGI-E) | 12, 24 and 52 weeks
  The patient global functioning will be assessed by means of the Clinical Global Impression (CGI) Scales. The Early Clinical Drug Evaluation Program (ECDEU) version of the CGI is a 3-item clinician rated scale that measures illness severity (CGI-S), global improvement or change (CGI-I) and treatment response (efficacy index: CGI-E).
  The CGI-E score should take account of both therapeutic effect and tolerance, and ranges from 0 (marked improvement and no toxicity) and 4 (unchanged or worse and toxicity outweigh the therapeutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.
  The calculation of the scores will be performed according to the instructions obtained from copyright holders.
Daytime Sleepiness | 12, 24 and 52 weeks
  Daytime Sleepiness will be assessed by means of the Epworth Sleepiness Scale (ESS). The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different daily activities. The ESS score can range from 0 to 24. The higher the ESS score, the higher that person Average Sleep Propensity in Daily Life (ASP), or their daytime sleepiness across a wide range of activities in their daily lives.
Hospital Anxiety and Depression | 12, 24 and 52 weeks
  Anxiety and depression symptoms will be assessed by means of the the Hospital Anxiety and Depression Scale (HADS). This is a patient self-reported instrument consisting of 14 items that provide scores on two specific subscales: "Anxiety" subscale (HADS-A, 7 items) and "Depression" subscale (HADS-D, 7 items).
  All items were scored on a 4-point Likert scale from 0 ("never") to 3 ("almost every day") referring to overt symptoms within the last week. Total scores range from 0 to 21 points for each subscale, with higher scores indicating higher levels of symptoms.
Retention with cenobamate | 52 weeks
  Retention with cenobamate will be assessed by calculating the frequency of patients still on treatment with cenobamate at 52 weeks of treatment initiation.

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Policlinico di Bari, Bari, Bari
  - Università degli Studi di Catanzaro "Magna Graecia", Catanzaro, Catanzaro
  - IRCCS Neuromed, Pozzilli, Isernia
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia, Pavia
  - Campus Bio-Medico, Roma, Roma
  - Policlinico Umberto I, Roma, Roma
  - Humanitas Gradenigo, Torino, Torino
  - Associazione La Nostra Famiglia - IRCCS Eugenio Medea, Conegliano, Treviso
  - Azienda Sanitaria Universitaria (A.O.U.) Integrata, Udine, Udine
  - Ospedale San Bortolo, Vicenza, Vicenza

REFERENCES:
- [Derived] Lattanzi S, Ranzato F, Di Bonaventura C, Bonanni P, Gambardella A, Tartara E, Assenza G, Procaccini M, Falsetto N, Villano V, Camattari G, Ori A, Di Gennaro G; BLESS Study Group. Effectiveness and Safety of Adjunctive Cenobamate in People with Focal-Onset Epilepsy: Evidence from the First Interim Analysis of the BLESS Study. Neurol Ther. 2024 Aug;13(4):1203-1217. doi: 10.1007/s40120-024-00634-5. Epub 2024 Jun 8. PMID 38850402